CLINICAL TRIAL: NCT05734781
Title: Development and Evaluation of a Culturally Specific End-of-life Communication Skills Training for Chinese Oncology Nurses
Brief Title: End-of-life Communication From a Chinese Perspective
Status: Completed | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Joyce Chung, Assistant Professor, School of Nursing, The Hong Kong Polytechnic University
Other Study IDs: HSEARS20221217002
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Terminally Ill
Keywords: Communication; Health personnel; Terminally ill; Adult
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Interviewees: terminally ill patients, families and healthcare providers of such patients
  Interventions: Other: Not Application as this is a qualitative study

INTERVENTIONS:
Other: Not Application as this is a qualitative study — Not Application as this is a qualitative study

SUMMARY:
The goal of this observational study is to explore experiences and perceptions of end-of-life communication in Chinese terminally ill patients, families and healthcare providers. The main question it aims to answer is:

• What are the experiences and perceptions of end-of-life communication in Chinese terminally ill patients, families and healthcare providers? Participants will be invited to either semi-structured in-depth interviews or focus group discussions to share their thoughts.

DETAILED DESCRIPTION:
Objectives: To explore stakeholders' (patients, families and healthcare providers) experiences and perceptions of end-of-life communication in China; and understand culturally appropriate communication strategies.

Design and subjects: This study is a qualitative study. Eligible patients, family caregivers and healthcare providers will be recruited in two hospitals. Purposive sampling methods will be adopted. Semi-structured in-depth interviews with patients and family caregivers will be conducted respectively. Focus group discussions will be arranged with healthcare providers, allowing them to discuss end-of-life communication and generate group interactions and creative thinking.

Data analysis: The data analysis will be an iterative, cyclic and self-reflective process. Using inductive thematic analysis, common themes and categories will be determined through inductive reasoning and constant comparison.

Expected results: The study will fill the gap of no empirical evidence on end-of-life communication strategies from a Chinese perspective and enrich the knowledge about end-of-life communication.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Be aged older than 18 years
* Have a defined incurable life-limiting illness with a likely life expectancy of fewer than 12 months (National Institute for Health and Care Excellence, 2021), according to the consultation with the patient's physician
* Have been informed of disease diagnosis and treatment
* Be able to speak Mandarin and express clearly
* Be able to provide informed consent

Family caregivers:

* Be aged older than 18 years
* One of the terminally ill patient's primary family caregivers who are familiar with patient's situation, which is defined as lived with or visited patients at least twice a week in the past month
* Have been informed of patient's disease diagnosis and treatment
* Be able to speak Mandarin
* Be able to provide informed consent

Healthcare providers:

* Be nurses, physicians or other healthcare professionals
* Be experienced in providing treatment or care to patients with advanced, life-limiting illnesses (whose likely life expectancies of fewer than 12 months) and family caregivers of such patients for at least five years (Koh et al., 2016)
* Consent to participate in the study

Exclusion Criteria:

Patients and family caregivers:

* Severe auditory impairment
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Terminally ill patients (whose likely life expectancies of fewer than 12 months), families and healthcare providers of such patients
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Qualitative data and participants basic information | Through study completion, an average of 12 months
  Interviews and focus group discussions will be conducted to collect qualitative data

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Chung, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen W, Chung JOK, Lam KKW, Molassiotis A. Patients', families' and healthcare providers' perspectives on end-of-life communication in Chinese hospital settings: A qualitative study protocol. PLoS One. 2023 Dec 27;18(12):e0296342. doi: 10.1371/journal.pone.0296342. eCollection 2023. PMID 38150444